CLINICAL TRIAL: NCT04517266
Title: Evaluating Omitting of Internal Mammary Irradiation Among Early Stage Intermediate Risk (N1) Breast Cancer Patients According to Clinical-genomic Model: an Open Label, Non-inferior Randomized Controlled Trial
Brief Title: Evaluating Omitting of Internal Mammary Irradiation Among Early Stage Intermediate Risk (N1) Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, QIWEIXIANG, Clinical Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020(55)
Record Dates: First submitted 2020-08-12; First posted 2020-08-18 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; N1; clinical-genomic model; genomic model; radiotherapy; internal mammary irradiation; clinical model
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): whole breast/chest wall irradiation + SVC irradiation
  Interventions: Radiation: omit of IMI group
- controlled group (Active Comparator): whole breast/chest wall irradiation + IMI+SVC irradiation
  Interventions: Radiation: IMI group

INTERVENTIONS:
Radiation: omit of IMI group — clincial high risk breast （≥2 risk factors）patients with 18-gene low risk an indication for regional nodal irradiation will received 2 Gy for 25 fractions to chest wall or whole breast and supraclavicular lymph nodes irradiation and sequential tumor bed boost of 2 Gy for 5 fractions following breast conserving surgery.
  Arms: experimental group
Radiation: IMI group — clincial high risk breast （≥2 risk factors）patients with 18-gene low risk an indication for regional nodal irradiation will received 2 Gy for 25 fractions to chest wall or whole breast and supraclavicular lymph nodes irradiation and sequential tumor bed boost of 2 Gy for 5 fractions following breast conserving surgery.
  Arms: controlled group

SUMMARY:
The effect of internal mammary irradiation (IMI) added to whole-breast or thoracic-wall irradiation plus supraclavicular (SVC) irradiation after surgery on survival among women with early-stage intermediate risk (N1) breast cancer remains debated. The present study aimed to identified patient could be omitted from internal mammary lymph node irradiation by using a clinical-genomic model.

DETAILED DESCRIPTION:
This study is a phase II open label, non-inferior randomized controlled trial, we aimed to compare the safety and effectiveness difference of whole breast/chest wall irradiation + IMI+SVC irradiation vs whole breast/chest wall irradiation + SVC irradiation among clinical high risk, genomic low risk of N1 breast cancer.

In previous studies, 28 gene classifier has been developed and established to predict local/regional recurrence. The 28 gene classifier was combined with 18 cancer gene and 10 reference gene. The 18 cancer gene includes BLM, TCF3, PIM1, RCHY1, PTI1,DDX39, BUB1B, STIL, TPX2, CCNB1,MMP15, CCR1,NFATC2IP, TRPV6,OBSL1, C16ORF7,DTX2, and ENSA. The expression of RCHY1, PTI1, ENSA, and TRPV6 is associated with better tumor biology and disease control. The remaining 14 genes are associated with poor outcomes. By using the 18-gene scoring algorithm defines the risk of recurrence as: low risk or high risk.

A total of five clinical factors [age（≤40 vs. >40, number of positive lymph node（1-2 vs. 3）, grade(I-II vs. III), tumor size (T1-T2), ki-67(<14% vs. ≥14%)] were identified to be significantly associated with outcomes of breast cancer in our previous study. And patients with more than 2 risk factors were defined as clinical high risk.

Clinical high risk participants (≥2 factors) with low-risk scores will be randomized to whole breast/chest wall irradiation + IMI+SVC irradiation or whole breast/chest wall irradiation + SVC irradiation

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed invasive breast cancer

  * Underwent radical surgery with either mastectomy or breast conserving surgery and axillary lymph node dissection (ALND)
  * The number of positive lymph node should be 1-3 (N1).
  * Clinical high risk breast cancer (≥2 clinical risk factors)
  * Aged 18-80 years old
  * ECOG performance status ≤2 (Karnofsky ≥70%) Anticipative overall survival >5 years Pathologically surgical margin >2mm ER (estrogen-receptor), PR (progesterone-receptor), HER2 (human epidermal growth factor receptor 2) and Ki67 testing can be performed on the primary breast tumor Women of child-bearing potential must agree to use adequate contraception for up to 1 month before study treatment and the duration of study participation Ability to understand and willingness to participate the research and sign the consent form

Exclusion Criteria:

* • Axillary dissection of less than 10 lymph nodes

  * Pathologically positive ipsilateral supraclavicular lymph node
  * Pathologically or radiologically confirmed involvement of ipsilateral internal mammary lymph nodes
  * Pregnant or lactating women
  * Treated with breast reconstruction surgery
  * Severe non-neoplastic medical comorbidities
  * History of non-breast malignancy within 5 years with the exception of lobular carcinoma in situ, basal cell carcinoma of the skin, carcinoma in situ of skin and carcinoma in situ of the cervix
  * simultaneous contralateral breast cancer
  * Previous radiotherapy to the neck, chest and/or ipsilateral axillary region
  * Active collagen vascular disease
  * Definitive pathological or radiologic evidence of distant metastatic disease
  * Primary T4 tumor
  * Interval between radical surgery (mastectomy or breast conserving surgery) and radiotherapy was more than 12 weeks or interval between last dose of adjuvant chemotherapy and radiotherapy was more than 8 weeks

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
2-year event-free survival | 2 years
  any recurrence,distant metastasis or death in 2 years

SECONDARY OUTCOMES:
5-year event-free survival | 5 years
  any local recurrence, distant metastasis or death in 5 years
5-year overall survival | 5 years
  death in 5 years
5-year Locoregional recurrence (LRR) | 5-years
  any first recurrence confirmed by histology or cytology within the ipsilateral chest wall and/or regional nodes area (including supraclavicular, infraclavicular or internal mammary lymph nodes)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Xiang Qi, Dr., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai jiaotong univestigy school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng SH, Horng CF, Huang TT, Huang ES, Tsou MH, Shi LS, Yu BL, Chen CM, Huang AT. An Eighteen-Gene Classifier Predicts Locoregional Recurrence in Post-Mastectomy Breast Cancer Patients. EBioMedicine. 2016 Feb 16;5:74-81. doi: 10.1016/j.ebiom.2016.02.022. eCollection 2016 Mar. PMID 27077114
- [Background] Cheng SH, Horng CF, West M, Huang E, Pittman J, Tsou MH, Dressman H, Chen CM, Tsai SY, Jian JJ, Liu MC, Nevins JR, Huang AT. Genomic prediction of locoregional recurrence after mastectomy in breast cancer. J Clin Oncol. 2006 Oct 1;24(28):4594-602. doi: 10.1200/JCO.2005.02.5676. PMID 17008701
- [Background] Qi WX, Cao L, Xu C, Zhao S, Chen J. Adjuvant regional nodal irradiation did not improve outcomes in T1-2N1 breast cancer after breast-conserving surgery: A propensity score matching analysis of BIG02/98 and BCIRG005 trials. Breast. 2020 Feb;49:165-170. doi: 10.1016/j.breast.2019.11.001. Epub 2019 Nov 29. PMID 31812892
- [Derived] Qi WX, Cao L, Zheng S, Xu C, Cai R, Xu H, Cai G, Chen J. IMNI PRECISION trial protocol: a phase II, open-label, non-inferior randomized controlled trial of tailoring omission of internal mammary node irradiation for early-stage breast cancer. BMC Cancer. 2022 Dec 27;22(1):1356. doi: 10.1186/s12885-022-10454-1. PMID 36575421